CLINICAL TRIAL: NCT00505297
Title: A Longitudinal Study of Osteoarthritis (OA) Disease Progression Measured by MRI, dGEMRIC, and Radiography
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: Pfizer (Industry)
Other Study IDs: A9001140; H6513-25393
Record Dates: First submitted 2007-07-20; First posted 2007-07-23 (Estimated); Last update posted 2007-07-23 (Estimated); Status verified 2006-10

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis (OA); Magnetic Resonance Imaging (MRI); delayed Gadolinium Enhanced MRI of cartilage (dGEMRIC); disease modifying osteoarthritis drug (DMOAD); Potentially rapidly progressing osteoarthritis; MRI measurement of cartilage
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- A: Subjects with potentiall rapidl progressing OA
- B: Age-matched healthy subjects with no knee pain

SUMMARY:
In order to design future disease modifying osteoarthritis drug (DMOAD) proof of concept studies, this study is being conducted to assess magnetic resonance imaging (MRI) measurements of cartilage morphology and glycosaminoglycan (GAG) content as it relates to the progression of disease in subjects with potentially rapidly progressing OA. The subject population is selected to have higher likelihood of having rapidly progressing OA (i.e., a more rapid joint space narrowing (JSN) compared to general knee OA population and thus, may be more likely to have changes in GAG content and/or cartilage volume. The results of this study may provide a reasonable means to assess DMOAD activity of drugs in development. The non-OA controls are included to determine the rate of change for subjects of similar age. Ideally, results of this study will identify reliable methods for delayed Gadolinium Enhanced MRI of cartilage (dGEMRIC) and MRI cartilage assessment that correlate with OA disease progression as compared to x-ray changes.

DETAILED DESCRIPTION:
The objective of the study are:

* Evaluate OA progression by evaluating cartilage morphology, cartilage glycosaminoglycan (GAG) content, and joint space changes measured by MRI (3.0T), dGEMRIC index, and radiography, respectively using age-matched control subjects to identify disease related changes.
* Identify subject characteristics associated with more rapidly progressing OA.
* Identify most sensitive efficacy endpoints for future DMOAD proof of concept (POC) studies.
* Establish time interval for future studies based on MRI endpoints.
* Evaluate the effect of contrast agent on MRI cartilage morphology and T2 measurements
* Define criteria for classifying cartilage legions/deficits using dGEMRIC and T2 measurements.
* Collect biofluid samples for future validation of disease specific biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Female patients evaluated to be relatively in good health
* 40 years old and above
* Negative pregnancy test

Additional inclusion criteria for OA patients:

* Frequent knee symptoms in the past year, defined as:
* pain, aching, or stiffness on most days of a month during the past year
* use od medication (all types) for treatment of knee pain on most days of a month during the past year
* Kellgren & Lawrence Grades 2 or 3 of the study knee (with either the same or less severe OA , or no OA in the contralateral knee)
* Body mass index (BMI) of 30 and above
* Medial joint space width of 2 mm and above

Additional inclusion criteria for age-matched controls:

* BMI of 28 and above
* No evidence of knee OA in either knee (i.e., Kellgren & Lawrence Grade 0 diagnosed by x-ray on AP view; infrequent knee pain, aching, stiffness during the past year; infrequent use of medication (all types) for treatment of knee pain during the past year.

Exclusion Criteria:

* Anticipated need for knee surgery in the next 2 years
* OA predominantly in the lateral tibiofemoral compartment measured by PA x-ray view of the study knee
* Intra-articular steroids to study joint (3 month washout), intra-articular hyaluronic acid to the study joint (3 month-washout), doxycycline (3 month washout), or arthroscopy within the last 6 months
* Medial joint space width less than 2 mm measured by PA view of knee x-ray
* History of joint replacement, intra-articular fracture, osteotomy, arthroplasty, or meniscectomy of the study knee
* History of other diseases that may involve the study joint including inflammatory joint diseases, crystalline disease, endocrinopathies, metabolic, diseases, knee infection of the study knee, neuropathic disorders, avascular necrosis, Paget's disease, or tumors (chondrocalcinosis is acceptable; treated thyroid disease is acceptable)
* Systemic inflammatory diseases (e.g., Rheumatoid arthritis)
* Other pain that the principal investigator feels can not be distinguished from knee pain (e.g., lumbar pain, hip pain, trochanteric bursitis)
* Musculoskeletal pain that may preclude the subject from remaining motionless for the MRI acquisitions
* Unable to undergo an MRI exam of the knee because of contraindications
* Unable to receive gadopentate contrast agent injection because of contraindications. A study subject who displays any sign of an allergic reaction to the contrast agent will be withdrawn from the dGEMRIC part of the protocol and will not receive any subsequent contrast agent injection. The subject may continue to complete the remainder fo the study, which includes MR morphometry scan, collection of blood and urine sample for biomarker assays, and completion of study questionnaires.
* Clinical chemistry laboratory values more than 2 times the upper limit of normal
* Participation in clinical trial with a study during in the past 14 days
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with trial participation or may interfere with the interpretation of trial results and, in the judgment of the investigator, would make the subject inappropriate for entry in the this trial

Min Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2004-08; Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharmila Majumdar, PhD, Principal Investigator — University of California, San Francisco; Thomas M. Link, M.D., Principal Investigator — University of California, San Francisco
Locations (1):
- University of California - San Frnacisco, San Francisco, California, United States